CLINICAL TRIAL: NCT04361656
Title: The Effect of Adding Lubiprostone to Standard Large-Volume PEG-ELS on The Quality of Inpatient Colonoscopy Preparation.
Status: Withdrawn | Type: Observational
Why Stopped: Endoscopy services were suspended in March 2019 due to COVID-19 pandemic. Study was not restarted.
Sponsor: Henry Ford Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 1474341
Record Dates: First submitted 2020-01-13; First posted 2020-04-24 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2022-03

CONDITIONS: Colonoscopy Preparation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Current standard of care preparation: Current Standard of Care for inpatient colonoscopy: The dose of PEG-ELS will be large-volume (4-Liter) administered as either single-dose if colonoscopy is scheduled BEFORE 11 a.m. (250 mL orally every 15 minutes between 6 p.m. and midnight the day prior to procedure), or split-dose if the colonoscopy is scheduled AT or AFTER 11 a.m. (First dose: 2-Liters; 250 mL orally every 15 minutes between 6-8 p.m. the day prior to procedure. Second dose: 2-Liters; 250 mL orally every 15 minutes to be completed 5 hours before the scheduled time of the procedure).
  Interventions: Drug: PEG-ELS current standard of care
- Lubiprostone Intervention: The study entails giving two doses of Lubiprostone in addition to the standard large-volume polythene glycol-electrolytes solution (PEG-ELS) according to the time of the procedure as follow: If the colonoscopy is scheduled BEFORE 11a.m. the patient will receive in addition to the PEG-ELS: Lubiprostone 24 mcg capsule orally (roughly every 12 hours) for total of 2 doses, with the last dose being at least 4 hours prior to the scheduled colonoscopy.
  If the colonoscopy is scheduled AT or AFTER 11a.m. the patient will receive in addition to PEG-ELS: Lubiprostone 24 mcg capsule orally 2 hours before each dose of the PEG-ELS
  Interventions: Drug: PEG-ELS current standard of care plus Lubiprostone 24 microgram Oral Cap (x2)

INTERVENTIONS:
Drug: PEG-ELS current standard of care — Standard of care for inpatient colonoscopy
  Groups: Current standard of care preparation
Drug: PEG-ELS current standard of care plus Lubiprostone 24 microgram Oral Cap (x2) — The dose of Lubiprostone will be 24 mcg capsule orally (roughly every 12 hours) for total of 2 doses, with the last dose being at least 4 hours prior to the scheduled colonoscopy if it is BEFORE 11 a.m., and Lubiprostone 24 mcg capsule orally 2 hours before each dose of the PEG-ELS if colonoscopy is scheduled AT or AFTER 11 a.m..
  Groups: Lubiprostone Intervention

SUMMARY:
This is a multicenter interrupted-time series study. The study will include patients between the age of 18-85 year old, both males and females, who are scheduled for inpatient colonoscopy procedure.

The study will be divided into two phases:

The initial phase will be a prospective review of inpatient colonoscopy procedure between September, 1st 2020 and March, 31st 2021 to assess overall adequacy of inpatient colonoscopy preparation and patient satisfaction at the three participating sites using standard of care colonoscopy preparation prior to implement our intervention.

The intervention phase will take place between April, 1st 2021 and October 31st 2021, where all patient undergoing inpatient colonoscopy procedures will receive Lubiprostone in addition to large-volume PEG-ELS.

The patients will be evaluated with colonoscopy the next day. The preparation quality will be documented using the Boston Bowel Preparation Scale (BBPS).

DETAILED DESCRIPTION:
2. INTRODUCTION AND BACKGROUND 2.1. Study rationale and aim An excellent bowel preparation is crucial to perform a high-quality colonoscopy and essential to visualize the entire colonic mucosa and to increase the safety of therapeutic maneuvers. Prior studies revealed that inpatient setting was associated with higher rate of poor bowel preparation which led to lower rate of procedure completion. The addition of Lubiprostone to standard PEG-ELS bowel preparation for colonoscopy was evaluated in the outpatient setting and revealed significantly better colon cleansing, decrease total length of procedure, and improved the overall patient satisfaction with the preparation.

The aim of this trial is to evaluate the effect of adding Lubiprostone to standard large-volume PEG-ELS on the bowel preparation for inpatient colonoscopy.

2.2. Background Colonoscopy is a procedure that permits direct visualization, examination and treatment of the rectum, colon and terminal ileum. It can be used for both diagnostic and therapeutic purposes. In order to perform a high-quality colonoscopy examination, the American Society of Gastrointestinal Endoscopy/American College of Gastroenterology Taskforce on Quality in Endoscopy committee established a pre-, intra- and post-procedural quality indicators. Bowel preparation is one of the most important pre-procedural indicators, as an excellent preparation is crucial to visualize the entire colonic mucosa and to increase the safety of therapeutic maneuvers. Multiple studies revealed rates of incomplete colonoscopy between 10-20%, Sidhu et al revealed a rate of 7.8% of incomplete colonoscopies with inadequate bowel preparation being the most common culprit. It has been reported that inadequate or poor preparation occurs in 20-25% of colonoscopies in the United States. The diagnostic yield, safety and quality indicators (adenoma detection rate, withdrawal time and cecal intubation rate) of colonoscopy can be inversely affected by inadequate or poor bowel preparation, as it can lead to: Increase procedural duration, cancel or repeat procedures, increase health costs, a potential increase in complications and increase probability of missing neoplastic lesions or adenomatous polyps (28-42% patients had adenomas on repeated exam within 3 years).

Factors that can be associated with inadequate or poor bowel preparation has been evaluated by researchers in order to improve this quality indicator. It has been shown that inadequate preparation is more likely in the following situations: Inpatient status, prior inadequate bowel preparation, advanced age, comorbidities (obesity, cirrhosis, stroke, dementia, and Parkinson's), language barrier, polypharmacy, late colonoscopy starting time and failure to follow preparation instructions. Ness et al and Almadi et al in their studies found that inpatient setting was associated with higher rate of poor bowel preparation which led to lower rate of procedure completion and terminal ileum intubation. An ideal bowel cleansing preparation should be safe, tolerable, affordable, and can reliably empty the colon in a timely fashion without altering the colonic mucosa histology. The large-volume polyethylene glycol-electrolyte solution (PEG-ELS) is one of the most used FDA approved bowel preparation methods. PEG-ELS is an inert polymer of ethylene oxide formulated as a non-absorbable solution which is osmotically balanced with non-fermentable electrolyte solutions. It passes through the gastrointestinal tract without net absorption, secretion, or significant effect on fluid and electrolyte shift. Giving part of the bowel preparation does on the same day as the colonoscopy (termed split-does) results in a higher quality colonoscopy examination compared with ingestion of the entire preparation on the day or evening before colonoscopy.

As no available preparation has all of the ideal characteristics, studies evaluated the effect of adding other medications to enhance the quality of the preparation. The routine addition of prokinetic agents or bisacodyl to one of the standard regimens (Polyethylene glycol-electrolyte solution) did not improve patient tolerance or colonic cleansing.

Lubiprostone is a derivative of prostaglandin E1 which has been shown to be effective in treating Chronic Idiopathic Constipation, Opioid Induced Constipation and Irritable Bowel Syndrome-Constipation (IBS-C). Lubiprostone works by stimulating and inducing the secretion of chloride by activating chloride channel Type-2 and cyctic fibrosis transmembrane conductance regulator chloride channels in the apical membrane of the intestinal epithelial cells. Ultimately, the release of chloride ions from the cells into the intestinal lumen results in increase fluidity within the lumen itself. Furthermore, the increase of fluid contents within the lumen results in increase luminal distention which promotes the gastrointestinal tract motility, resulting in an increase in intestinal and colonic transit. By increasing the fluid content within the luminal wall and increasing intestinal and colonic transit, the resultant benefit is softening of stool and rather rapid and facilitated emptying of colonic contents which results in improvement in constipation and efficient colonic emptying.

Joel et al, and Banerjee et al evaluated the addition of Lubiprostone to standard PEG-ELS bowel preparation for colonoscopy performed in the outpatient setting. They showed significantly better colon cleansing, decreased total length of procedure, and improved overall patient satisfaction with the preparation. Grigg et al revealed a trend toward improved quality of colonoscopy preparation by adding two doses of Lubiprostone to standard PEG in diabetic patients undergoing outpatient screening colonoscopy. Documentation of quality of bowel preparation is an important post-procedural quality indicator. The Boston Bowel Preparation Scale is one of the most commonly used validated systems in the literature for documentation of the colonoscopy preparation. It is a 10-point (0-9) summation score assessing bowel preparation quality in 3 segments of the colon after all cleansing maneuvers during colonoscopy.

2.3. Risk/Benefit assessment 2.3.1. Known potential risks Lubiprostone is an approved and licensed medication. The Product/Safety Information published on the company website (https://www.amitiza.com/hcp/safety-indication/chronic-idiopathic-constipation) was used as the primary source of the potential risks associated with Lubiprostone use.

"Lubiprostone is not for everyone". It is contraindicated in patients with known or suspected mechanical gastrointestinal obstruction. It should be avoided in patients with severe diarrhea and during pregnancy (unless the potential benefit justifies the potential risk to the fetus). Caution should be exercised when it is administered to a nursing woman. These were included as exclusion criteria. Syncope, hypotension and dyspnea have been reported within an hour of the first dose or subsequent doses of Lubiprostone and generally resolve prior to the next dose, but may recur with repeat dosing. In clinical trials of Lubiprostone (24 microgram (mcg) twice daily vs placebo), the most common adverse reactions (incidence > 4%) were nausea (29% vs 3%), diarrhea (12% vs 1%), headache (11% vs 5%), abdominal pain (8% vs 3%), abdominal distension (6% vs 2%), and flatulence (6% vs 2%). There was no clinically significant changes in serum electrolyte levels in adult patients with CIC receiving Lubiprostone.

Other potential risks associated with PEG-ELS and colonoscopy procedure are not included in this study protocol as they are considered part of the standard of care required for patient evaluation and not part of this research study.

2.3.2. Known potential benefits The addition of Lubiprostone to standard PEG-ELS bowel preparation for colonoscopy was evaluated in the outpatient setting and revealed significantly better colon cleansing, decrease total length of procedure, and improved the overall patient satisfaction with the preparation. This would potentially result in reduce health costs, decrease complications rate and enhance the accuracy of neoplastic lesions or adenomatous polyp detection rates.

3 STUDY OBJECTIVES AND OUTCOMES 3.1 Objectives 3.1.1 Primary objective The primary objective of this trial is to evaluate the effect of adding Lubiprostone to standard large-volume PEG-ELS on the bowel preparation for inpatient colonoscopy.

3.1.2 Secondary objectives

The secondary objectives of this trial are:

1. To determine the adverse events related to the addition of Lubiprostone to large-volume PEG-ELS.
2. To determine the overall patient satisfaction with the bowel preparation regimen with the addition of Lubiprostone to large-volume PEG-ELS.

ELIGIBILITY:
Inclusion Criteria:

* Is scheduled for colonoscopy evaluation during his hospitalization to one of the trial sites (SJPH, PPH, or SJMH).
* Has a negative urine pregnancy test (hCG) for female of reproductive age.
* Provide an Informed Consent / has a legally acceptable representative capable of understanding the Informed Consent document and providing consent on the participant's behalf.
* Provide a separate signed and dated Informed Consents for colonoscopy procedure and anaesthesia administration as per site policy.

Exclusion Criteria:

* Has a documented or suspected bowel obstruction (small bowel obstruction, volvulus, gastric outlet obstruction, ileus, or toxic megacolon).
* Has a documented gastroparesis.
* Has severe diarrhea (>8 bowel movements per day).
* Has severe encephalopathy or obtunded (GCS < 13).
* Has a documented or suspected acute coronary syndrome or recent myocardial infarction within 12 weeks prior to enrollment.
* Has renal impairment with GFR less than 30 ml/min/1.73 m2 on the day of enrollment (end-stage renal disease on renal replacement therapy can be enrolled).
* Has severe liver impairment with Child-Pugh class B or C.
* Has symptomatic heart failure (NYHA class III or IV) or prohibitive pre-procedure cardiac risk (documented by primary team or cardiology prior to enrollment).
* Has a known hypersensitivity to Lubiprostone or its class.
* Is pregnant or lactating.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital patients having colonoscopy performed
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-02-04 (Actual); Study Completion 2021-02-04 (Actual)

PRIMARY OUTCOMES:
Independent gastroenterologists BBPS review | scored at completion of all data collection,or after 2023
  The Boston Bowel Preparation Scale (BBPS) is a four-point scoring system (0-3) applied to each of the three broad regions of the colon: the right colon (including the cecum and ascending colon), the transverse colon (including the hepatic and splenic flexures), and the left colon (including the descending colon, sigmoid colon, and rectum). Scores can range from 0-9.
Participant satisfaction through standardized questionnaire form | 3 years
  Adverse symptoms following colonoscopy can range from none (0) to severe (4)

SECONDARY OUTCOMES:
Colonoscopy procedure BBPS by performing gastroenterologist | 3 years
  The Boston Bowel Preparation Scale (BBPS) is a four-point scoring system (0-3) applied to each of the three broad regions of the colon: the right colon (including the cecum and ascending colon), the transverse colon (including the hepatic and splenic flexures), and the left colon (including the descending colon, sigmoid colon, and rectum). Scores can range from 0-9.
Adverse event reporting | 3 years
  any EHR documented adverse event during current hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zakaria, MD, Principal Investigator — Henry Ford Health System
Locations (3):
- United States (3):
  - Ascension Providence Hopsital (Novi), Novi, Michigan
  - Ascension Providence Hospital, Southfield Campus, Southfield, Michigan
  - Ascension Macomb-Oakland Hospital, Warren, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grigg E, Schubert MC, Hall J, Rahhal F, Raina D, Sridhar S, Chamberlain SM. Lubiprostone used with polyethylene glycol in diabetic patients enhances colonoscopy preparation quality. World J Gastrointest Endosc. 2010 Jul 16;2(7):263-7. doi: 10.4253/wjge.v2.i7.263. PMID 21160617